CLINICAL TRIAL: NCT03275246
Title: Establish Implant Accuracy With X-PSI Knee System - A Multi-center, Prospective, Non-controlled Post Market Study
Brief Title: Establish Implant Accuracy With X-PSI Knee System
Acronym: X-PSI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical study was stopped due to very low enrolment numbers. Due to the very slow enrolment, the goal of the study cannot be reached within a reasonable time frame.
Sponsor: Zimmer, GmbH (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSE2017-01K
Record Dates: First submitted 2017-08-24; First posted 2017-09-07 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis; Post-traumatic Osteoarthritis
Keywords: Primary total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total knee arthroplasty (Experimental): Patients undergoing total knee arthroplasty
  Interventions: Device: X-PSI Knee System

INTERVENTIONS:
Device: X-PSI Knee System — Patients are operated with X-PSI Knee System guides

SUMMARY:
The goal of this study is to establish the accuracy of the new X-PSI Knee System guides by analyzing early postoperative (4-6 weeks) imaging data with regards to the mechanical alignment and compare them with preoperative planning imaging data. Mechanical alignment in the hip-knee-ankle (HKA) frontal plane with X-PSI Knee System will be measured and compared with results reported in the literature using a conventional (non-guided) approach.

Hypothesis: The use of the new X-PSI Knee System achieves the same accuracy with respect to mechanical alignment as with conventional instrumentation.

DETAILED DESCRIPTION:
Patient-specific instruments (PSI) provide surgeons with an anatomically personalized surgery tool. The newly developed and CE-marked X-PSI Knee System is based on long leg x-rays that are used to generate a pre-operative 3D model of the knee. The total knee replacement surgery will be planned according to this 3D model.

The aim of this multi-center, prospective, non-controlled post-market study is to scientifically document the accuracy, cost-effectiveness and subsequent clinical performance of the X-PSI Knee System. The X-PSI pin guides are designed to facilitate a more simplified, efficient and customized TKA procedure compared to conventional, non-guided instrumentation.

To evaluate the accuracy of the X-PSI Knee System, early postoperative (4-6 weeks) imaging data will be analysed with regards to the mechanical alignment (hip-knee-ankle angle) of the leg and matched to preoperative planning imaging data. The X-PSI Knee System cohort will then be compared with current literature (70% of cases within ±3 degrees) where patients were conventionally operated with non-guided surgery. No control group will be studied.

The cost-effectiveness of the X-PSI Knee System will be evaluated with an efficiency matrix to record OR set-up time, surgery time and post-processing time.

Clinical outcome data of the patients will be evaluated 4-6 weeks and 1 year post-surgery with the help of patient questionnaires (VAS pain scale, EQ-5D and Oxford Knee Score), a physical exam and the assessment of radiographs.

The study population will be compromised of males and females requiring total knee arthroplasty and satisfy the inclusion/exclusion criteria. The study will last one (1) year from the time of surgery. The collected data aim to improve the treatment and quality of life of patients suffering from degenerative joint diseases. In addition, shorter surgery times possibly result in reduced risk of infection, decreased time of anaesthesia and better cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient can follow the X-PSI Knee System imaging protocol as part of standard of care procedures.
* Patient gets TKA treatment which follows the criteria of the appropriate Instruction for Use.
* Patient is willing and able to cooperate in the required postoperative standard of care.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the study-related Informed Consent process and has signed the Ethics Committee approved Informed Consent

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient meets exclusion criteria of the appropriate Instruction for Use
* Patients who have any condition which would in the judgement of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, or is a known drug abuser, a known alcoholic or anyone who cannot understand what is required from them
* Patient is known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Schaetti, PhD, Study Chair — Jr. Clinical Project Lead
Locations (4):
- Germany (2):
  - HELIOS Kliniken Mittelweser GmbH, Nienburg
  - Knie Praxis Prof. Dr. Tibesku, Straubing
- Zuyderland Medical Park, Sittard, Netherlands
- Royal Bournemouth Hospital, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Knee Arthroplasty
Started | 8
Completed | 2
Not Completed | 6
Not completed — Protocol Violation | 5
Not completed — The study was stopped before the patient reached the final 1 year follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline data collected and reported for those participants that underwent surgery with X-PSI Knee System
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 3

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Leg Alignment
Description: Achievement of mechanical leg alignment in HKA frontal plane (± 3 degrees) with X-PSI Knee System is as accurate as with standard instrumentation at 4-6 weeks post operation. The X-PSI Knee System cohort will be compared with current literature (70% of cases within ± 3 degrees). No control group will be studied.
Time Frame: 4-6 weeks post-surgery
Population: Mechanical alignment data were not collected from any participant.
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 0

2. Secondary Outcome: Cost-effectiveness of the X-PSI Knee System Using an Efficiency Matrix
Description: The cost-effectiveness of the X-PSI Knee System will be measured using an efficiency matrix where OR set-up time, surgery time and tray sterilization times will be collected and compared to conventional TKA procedures.
Time Frame: During surgery, immediate pre- and post-surgery processing time
Population: No data on cost-effectiveness and efficiency were collected from any participant.
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Patient Clinical Outcome Measure: Visual Analog Score Pain
Description: Obtain clincal outcome data on patients treated using the X-PSI Knee System in primary TKA procedures. The pain level will be measured using a 10 cm long scale indicating no pain (0) and worst imaginable pain (10).
Time Frame: Baseline, 4-6 weeks and 1 year post-surgery
Population: Data should be interpreted with caution, as too few participants were followed to assess endpoints (N=3 for baseline and 4-6 weeks; N=2 for 1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 3
units on a scale
  Baseline | 8.2 (0.9)
  4-6 weeks post-surgery | 3.7 (2.4)
  1 year post-surgery: number analyzed (Participants) | 2
  1 year post-surgery | 1.1 (0.4)

4. Other Pre Specified Outcome: Patient Clinical Outcome Measure: Oxford Knee Score
Description: The Oxford Knee Score (OKS) is a 12-item patient-reported patient reported outcome specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). The OKS provides a single summed score which reflects the severity of problems that the respondent has with their knee. Each question (item) is scored from 0 to 4 with 0 being the worst outcome and 4 being the best outcome. The scores are then summed to produce an overall score running from 0 (worst possible) to 48 (best outcome).
Time Frame: Baseline, 4-6 weeks and 1 year post-surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 3
score on a scale
  Baseline | 18.3 (6.6)
  4-6 weeks post-surgery | 30.3 (5.3)
  1 year post-surgery: number analyzed (Participants) | 2
  1 year post-surgery | 45.0 (2.0)

5. Other Pre Specified Outcome: Patient Clinical Outcome Measure: EQ-5D Visual Analogue Scale (VAS)
Description: Obtain clincal outcome data on patients treated using the X-PSI Knee System in primary TKA procedures. The EQ-5D VAS is a score to measure general quality of life. The general health state will be assessed on a patient self-reported Visual Analog Scale (VAS) where the endpoints are labelled 0 (worst imaginable health state) to 100 (best imaginable health state). The VAS is used as a quantitative measure of health outcome that reflects the patient's own judgement.
Time Frame: Baseline, 4-6 weeks and 1 year post-surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 3
score on a scale
  Baseline | 73.3 (24.9)
  4-6 weeks post-surgery | 63.3 (12.5)
  1 year post-surgery: number analyzed (Participants) | 2
  1 year post-surgery | 91.5 (3.5)

6. Other Pre Specified Outcome: Patient Clinical Outcome Measure: EQ-5D-3L Descriptive System
Description: The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Time Frame: Baseline, 4-6 weeks and 1 year post-surgery
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 3
participants
  Baseline - patients reprting any problem (i.e some problems/ extreme problems) : Mobility | 2
  Baseline - patients reprting any problem (i.e some problems/ extreme problems) : Self-Care | 1
  Baseline - patients reprting any problem (i.e some problems/ extreme problems) : Usual Activities | 2
  Baseline - patients reprting any problem (i.e some problems/ extreme problems) : Pain/Discomfort | 3
  Baseline - patients reprting any problem (i.e some problems/ extreme problems) : Anxiety | 1
  4- weeks post-surgery patients reprting any problem (i.e some problems/ extreme problems) : Mobility | 2
  4- wks post-OP patients reprting any problem (i.e some problems/ extreme problems) : Self-Care | 0
  4- wks post-OP patients reprting any problem (i.e some problems/ extreme problems): Usual Activities | 2
  4- wks post-OP patients reprting any problem (i.e some problems/ extreme problems) : Pain/Discomfort | 3
  4- wks post-OP patients reprting any problem (i.e some problems/ extreme problems) : Anxiety | 2
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems) : Mobility: number analyzed (Participants) | 2
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems) : Mobility | 0
  1 year post-surgery patients reprting any problem (i.e some problems/ extreme problems) : Self-Care: number analyzed (Participants) | 2
  1 year post-surgery patients reprting any problem (i.e some problems/ extreme problems) : Self-Care | 0
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems): Usual Activities: number analyzed (Participants) | 2
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems): Usual Activities | 0
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems) : Pain/Discomfort: number analyzed (Participants) | 2
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems) : Pain/Discomfort | 1
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems) : Anxiety: number analyzed (Participants) | 2
  1 year post-OP patients reprting any problem (i.e some problems/ extreme problems) : Anxiety | 0

ADVERSE EVENTS:
Time Frame: 1 year starting from day of surgery
Description: Adverse Event data collected and reported for those participants that underwent surgery with X-PSI Knee System
Arm/Group | Total Knee Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to slow enrloment. Only 3 subjects were operated with X-PSI. Out of the 3 subjects, 2 reached the final 1 year follow-up. Due to the very low number of subjects, no statistical analysis was conducted on the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT03275246/Prot_SAP_000.pdf